CLINICAL TRIAL: NCT05509998
Title: Early Stage Identification and Engagement to Reduce the Duration of Untreated Psychosis: Evaluating the Impact of Screening and Systematic Communication
Brief Title: Reducing the Duration of Untreated Psychosis in the United States: The Impact of Screening and Systematic Communication
Acronym: EaSIE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yulia Landa, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 21-1631; 1R01MH130354-01 (NIH)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: First Episode Psychosis (FEP); Clinical High Risk for Psychosis (CHR)
Keywords: Duration of Untreated Psychosis (DUP); Screening; Communication; First Episode Psychosis (FEP); Clinical High Risk for Psychosis (CHR); Coordinated Specialty Care
MeSH Terms: conditions — Communication | interventions — High-Throughput Screening Assays; Mass Screening

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screening Method (SM) (Active Comparator): In the SM condition all consecutive incoming patients ages 12-30 entering mental health services will complete a self-report screener, the PQ-B on intake. The intake clinician will review the PQ-B and refer all patients who endorse 6 or more items for evaluation with the SIPS to determine whether the patient meets criteria for psychosis, CHR, or neither. Evaluating clinicians will meet with patients to discuss findings and make referrals to specialty care as appropriate. The evaluating clinician will follow-up with patients referred to CSC and CHR programs to determine date of initial engagement. This information will be corroborated with records from CHR and FEP programs.
  Interventions: Behavioral: Screening Method (SM)
- Screening and Communication Method (SCM) (Experimental): In the SCM condition, the same screening and evaluation procedures described above will continue, but clinicians conducting evaluations and making referrals will be trained to discuss findings and provide referrals using the ComPsych model. Following the evaluation, the clinician who conducted the evaluation will schedule a session with the patient, their family, and their treatment team (as applicable) and use the ComPsych model to discuss the findings of the evaluation, provide psychoeducation, and make referrals to specialty FEP or CHR services, as appropriate. The evaluating clinician will follow-up with patients referred to CSC and CHR programs to determine date of initial engagement. This information will be corroborated with records from CHR and FEP programs.
  Interventions: Behavioral: Screening and Communication Method (SCM)

INTERVENTIONS:
Behavioral: Screening Method (SM) — All consecutive incoming patients ages 12-30 entering mental health services will complete a self-report screener, the PQ-B on intake. The intake clinician will review the PQ-B and refer all patients who endorse 6 or more items for evaluation with the SIPS to determine whether the patient meets criteria for psychosis, CHR, or neither. Evaluating clinicians will meet with patients to discuss findings and make referrals to specialty care as appropriate.
  Arms: Screening Method (SM)
Behavioral: Screening and Communication Method (SCM) — Clinicians will be trained to discuss findings and provide referrals using the ComPsych model. ComPsych prepares clinicians to effectively communicate diagnostic, prognostic and treatment information about FEP and CHR with patients and families, using a model that instils realistic hope and provides information effectively to encourage shared decision making about treatment. All consecutive patients ages 12-30 entering mental health services will complete a self-report screener, the PQ-B on intake. The intake clinician will review the PQ-B and refer all patients who endorse 6 or more items for evaluation with the SIPS to determine whether the patient meets criteria for psychosis, CHR, or neither. Following the evaluation, the clinician will schedule a session with the patient, their family, and their treatment team (as applicable) and use the ComPsych model to discuss the findings of the evaluation, provide psychoeducation, and make referrals to specialty services, as appropriate.
  Arms: Screening and Communication Method (SCM)

SUMMARY:
The goal of this project is to investigate whether a systematic screening approach enhanced by an innovative model of communicating information about psychosis and treatment options to patients and families (ComPsych) can reduce Duration of Untreated Psychosis (DUP) by facilitating early identification of first episode psychosis (FEP) cases, rapid referral to specialty care and engagement in treatment. The study team will use a stepped-wedge cluster randomized controlled trial design to compare a systematic screening and communication method (SCM) to systematic screening method (SM) to evaluate whether SCM substantially reduces DUP. The study team hypothesize that: (1) SCM will result in a higher number of individuals initiating specialty services compared to SM; (2) The mean DUP of FEP individuals in SCM condition will be lower than the mean DUP of FEP individuals in SM condition, due to the reduced time to initiate FEP services. We will also conduct a qualitative study to examine implementation barriers and facilitators of SCM.

DETAILED DESCRIPTION:
Studies find a substantial delay between the onset of psychosis and the initiation of specialty treatment for first episode psychosis (FEP), with the duration of untreated psychosis (DUP) typically over one year in the U.S. Better strategies are needed to improve identification of individuals with FEP and to rapidly engage them in Coordinated Specialty Care (CSC) aimed at restoring functioning. This study will investigate whether a U.S. adaptation of a successful detection approach from the Netherlands enhanced by an innovative model of communicating information about psychosis and treatment options to patients and families (ComPsych), can reduce DUP. Researchers in the Netherlands compared screening of a consecutive help-seeking population entering mental health services to clinician referral from mental health clinics and found that screening captured significantly more individuals at clinical high risk for psychosis (CHR) and with FEP. Based on the Dutch model, within the Mount Sinai Health System in New York, the study team has piloted and established the feasibility of screening help-seeking youth entering mental health services with the aim of improving early identification of FEP cases and rapid referral to specialty care (Early Stage Identification and Engagement to Reduce DUP study (EaSIE), supported by NIMH R34). Individuals entering services are screened with the Prodromal Questionnaire-Brief Version (PQ-B). Those who screen positive are assessed by Structured Interview for Psychosis Risk Syndromes (SIPS) and referred to stage-specific specialty care (FEP or CHR services). To facilitate service engagement the study team developed, piloted, and established feasibility of the ComPsych model, a standardized training program for clinicians in delivering information about schizophrenia, psychosis and CHR to patients and families. The ComPsych model was developed based on qualitative studies with multiple stakeholders, which have shown that family involvement and clear communication about diagnosis are critical components to successful engagement in treatment and adherence to treatment recommendations. ComPsych aims to convey sensitive information in a way that promotes understanding, empathy, and a sense of ongoing support.

The objective of this project is to investigate whether a systematic screening approach enhanced by ComPsych can reduce Duration of Untreated Psychosis (DUP) by facilitating early identification of first episode psychosis (FEP) cases, rapid referral to specialty care and engagement in treatment. This study will use a Hybrid Type 1 randomized controlled trial design (RCT) to test the effectiveness of SCM vs SM and to examine multi-level implementation factors that can inform the identification of implementation strategies for future deployment of SCM in routine practice. This study team will use a stepped-wedge cluster RCT design to compare SCM to SM to evaluate whether SCM substantially reduces DUP. The study hypotheses are: (1) SCM will result in a higher number of individuals initiating specialty services compared to SM; (2) The mean DUP of FEP individuals in SCM condition will be lower than the mean DUP of FEP individuals in SM condition, due to the reduced time to initiate FEP services; (3) ComPsych targets (understanding of psychosis, stigma, attitudes about treatment) will mediate the impact of SCM on DUP. The study team will also conduct a multi-level qualitative implementation study informed by the Consolidated Framework for Implementation Research (CFIR) to first examine implementation barriers and facilitators and then apply the Expert Recommendations for Implementing Change (ERIC) taxonomy of implementation strategies to these findings to help select potential implementation strategies for SCM and SM. Data will be collected from clinicians and administrators before the implementation of the trial (year 1) and after recruitment for the trial has ended (year 4), and from patients and families throughout the project.

The knowledge gathered from this project is of significant public health relevance as it has potential to facilitate more rapid and timely detection and treatment of first episode psychosis (FEP) by evaluating the utility of systematic screening and communication strategies for psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age 12- 30
* ability to participate in assessments in English or Spanish
* ability to provide informed consent (assent for those under age 18)

Exclusion Criteria:

* previous diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or delusional disorder.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 912 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Duration of untreated psychosis (DUP) | up to 2 years
  The DUP is defined as the time, in weeks, between onset of psychotic symptoms (measured by the Symptom Onset in Schizophrenia Scale) and initiation of FEP treatment (date of intake into Coordinated Specialty Care (CSC) programs for first episode psychosis.

SECONDARY OUTCOMES:
Duration of unrecognized illness (DUI) | Baseline
  The DUI is defined as the time, in weeks, between onset of psychotic symptoms (measured by the Symptom Onset in Schizophrenia Scale) and evaluation with the SIPS.
Number of individuals initiating FEP services | up to 4 years
  Number of individuals initiating FEP services
Number of individuals initiating CHR services | up to 4 years
  Number of individuals initiating CHR services
Patient Satisfaction with Consultation Questionnaire (PSC) | Month 1
  This 22-item measure uses a 5-point Likert scale to measure satisfaction with amount/quality of information presented, emotional support and level of patient and family participation. The PSC has high internal reliability (Cronbach's Alpha .91). Used extensively in cancer studies, it is sensitive to differences in consultant behavior. For the purposes of this study, 4 items were removed. PSC will be administered to patients and family members in both SCM and SM conditions after a consultation where SIPS feedback is provided and referral made (in SCM ComPsych model will be used).
  Full scale from 18 - 90, with higher score indicating greater satisfaction
Knowledge About Schizophrenia Test (KAST) | Month 1
  A self-report scale adapted from the Knowledge About Schizophrenia Test (KAST) to assess understanding of psychosis. KAST is an 18 item instrument, full scale range from 1-18, higher score indicates more knowledge.
Stigma Scale (SS) | Month 1
  28-item Stigma Scale (SS) Full scale from 28 - 140, higher score indicates higher impact of stigma
Attitudes about treatment | Month 1
  Patients will be asked how much they agree (on a 5-point likert scale) with the statement: "I intend to go to my initial appointment at [name of program referred to]" Score from 1-5, with higher score indicating more agreement.
Attitudes about treatment | Month 1
  Patients will be asked how much they agree (on a 5-point likert scale) with the statement: "I think [program] is likely to help me with my problems". Score from 1-5, with higher score indicating more agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Landa, PsyD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH policy, a de-identified dataset will be uploaded to the NIMH Data Archive: the National Database for Clinical Trials Related to Mental Illness.